CLINICAL TRIAL: NCT01123278
Title: Testosterone Replacement in Metabolic Syndrome and Inflammation of Fat Tissue
Brief Title: Testosterone Replacement in Metabolic Syndrome and Inflammation
Acronym: TERMSINFAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Professor of Endocrinology, University of Roma La Sapienza
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TestoMet05
Record Dates: First submitted 2010-05-10; First posted 2010-05-14 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Hypogonadism; Metabolic Syndrome; Obesity; Erectile Dysfunction
Keywords: Adiponectin; Resistin; Adipocytes; Testosterone; Aging; HOMA-IR; Insulin; Hypogonadism; Metabolic Syndrome; Obesity; Erectile Dysfunction
MeSH Terms: conditions — Hypogonadism; Metabolic Syndrome; Obesity; Erectile Dysfunction; Insulin Resistance | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone gel (Experimental): Testosterone transdermal gel 50 mg/day
  Interventions: Drug: Testosterone
- Placebo gel (Placebo Comparator): Placebo gel
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone — Testosterone transdermal gel 50 mg/day (5 gr)
  Other Names: Androgel; Testogel
  Arms: Testosterone gel
Drug: Placebo — Placebo transdermal gel (5 gr)
  Arms: Placebo gel

SUMMARY:
Hypogonadism (HG) frequently complicates the Metabolic Syndrome (MetS), whether testosterone replacement (TRT) is beneficial has not been clearly ascertained. This study was designed to address the effects of TRT on insulin resistance, body composition and pro-inflammatory status in naïve patients with MetS and HG.

DETAILED DESCRIPTION:
The features of Metabolic Syndrome (MetS) include abdominal obesity, atherogenic dyslipidemia, raised blood pressure, insulin resistance or glucose intolerance. These symptoms are also frequently found in hypogonadal men.

Adipose tissue and androgens in male obesity are reciprocally linked. Total and free testosterone (T) are decreased in proportion to the degree of body fatness while T regulates insulin sensitivity and body composition. As a consequence, hypoandrogenism carries an additional independent risk for cardiovascular and metabolic disorders. Men with type 2 diabetes mellitus (T2D) exhibit lowered T levels that are inversely correlated to HbA1c. In addition, abdominal adiposity causes an impairment of testicular steroidogenesis that is directly linked to circulating adipokines; enhanced cytokine release from macrophage-infiltrated adipose tissue is pivotal to the pathogenesis of insulin resistance and atherosclerosis. Both MetS and T2D share with hypogonadism such a proinflammatory state.

For this reason we performed a randomized controlled trial on the effects of TRT on insulin resistance and circulating inflammatory markers in a cohort of middle-aged men with mild hypogonadism and MetS at first diagnosis, that were not taking medications known to influence the investigated outcomes. We established strict criteria for enrollment and used a physiological replacing therapy.

Given that testosterone replacement therapy (TRT) determines a reduction of body fat mass paralleled by an increase in fat free mass (6), and that TRT exerts an anti-inflammatory role inhibiting interleukins (IL), in particular the IL-6 gene (14), it remains to be established whether these independent effects also reflect in an improvement in insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* patients with Metabolic Syndrome according to ATPIII
* patients with mild hypogonadism (both testosterone evaluations between 6 and 11 nmol/L)
* patients naïve to hypoglycemic therapies

Exclusion Criteria:

* patients on hypoglycemic medications
* patients with severe hypogonadism (<5 nmol/L)
* patients with borderline T values hypogonadism (>11 nmol/L)
* patients with contraindication to testosterone therapy: prostate cancer, PSA>4 ng/ml, severe hepatic or renal insufficiency, Hb>17, Htc>52%, severe urinary retention

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2004-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Fat-Free Mass (kg) | 3 months
  Estimate of within subject absolute change in fat-free mass measured by DEXA (dual energy x-ray absorptiometry) at 3 months (90 days) interval during active or placebo treatment.

SECONDARY OUTCOMES:
Fat Mass (kg) | 3 months
  Estimate of within subject absolute change (Kg) in fat mass measured by DEXA at 3 months (90 days) interval during active or placebo treatment.
HOMA-IR (homeostasis model assessment)- (insulin resistance) | 3 months
  Estimate of within subject absolute change in measure of insulin resistance homeostatic model HOMA-IR.
CRP (C reactive protein) | 3 months
  C reactive protein (High sensitivity).
Interleukins | 3 months
  Within subject absolute and percentage change in serum:
  IL-1, IL-6, IL-10, IL-12, IL-2, IL-8, TNFa (tumor necrosis factor alpha)
Adipokines | 3 months
  Estimate of within subject absolute change in serum:
  ADIPONECTIN, LEPTIN, RESISTIN.
Waist circumference | 3 months
  Waist circumference (cm)
IIEF | 3 months
  International Index of Erectile Dysfunction
Penile CDU (color Doppler ultrasound) | 3 months
  Penile Color-Doppler Ultrasonography of cavernosal arteries before and after active or placebo treatment.
PSA (prostatic specific antigen) | 3 months
  PSA
Hb, Htc | 3 months
  haemoglobin and haematocrit
Fat-free mass | 6 months
Fat Mass | 6 months
HOMA-IR | 6 months
CRP | 6 months
Interleukins | 6 months
  Serum IL-1, IL-6, IL-10, IL-12, IL-2, IL-8, TNFa
Adipokines | 6 months
  Serum ADIPONECTIN, LEPTIN, RESISTIN.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Bonifacio, MD, PhD, Principal Investigator — University of Roma La Sapienza; Andrea M Isidori, MD, PhD, Study Director — University of Roma La Sapienza; Andrea Lenzi, MD, PhD, Study Chair — University of Roma La Sapienza
Locations (2):
- Italy (2):
  - Policlinico Umberto I Hospital - Sapienza University, Rome, Rome
  - Dipartimento di Fisiopatologia Medica - Policlinico Umberto I, Rome

REFERENCES:
- [Background] Isidori AM, Caprio M, Strollo F, Moretti C, Frajese G, Isidori A, Fabbri A. Leptin and androgens in male obesity: evidence for leptin contribution to reduced androgen levels. J Clin Endocrinol Metab. 1999 Oct;84(10):3673-80. doi: 10.1210/jcem.84.10.6082. PMID 10523013
- [Background] Aversa A, Isidori AM, Greco EA, Giannetta E, Gianfrilli D, Spera E, Fabbri A. Hormonal supplementation and erectile dysfunction. Eur Urol. 2004 May;45(5):535-8. doi: 10.1016/j.eururo.2004.01.005. PMID 15082192
- [Background] Isidori AM, Giannetta E, Pozza C, Bonifacio V, Isidori A. Androgens, cardiovascular disease and osteoporosis. J Endocrinol Invest. 2005;28(10 Suppl):73-9. PMID 16550728
- [Background] Isidori AM, Greco EA, Aversa A. Androgen deficiency and hormone-replacement therapy. BJU Int. 2005 Aug;96(2):212-6. doi: 10.1111/j.1464-410X.2005.05603.x. No abstract available. PMID 16001962
- [Background] Isidori AM, Giannetta E, Greco EA, Gianfrilli D, Bonifacio V, Isidori A, Lenzi A, Fabbri A. Effects of testosterone on body composition, bone metabolism and serum lipid profile in middle-aged men: a meta-analysis. Clin Endocrinol (Oxf). 2005 Sep;63(3):280-93. doi: 10.1111/j.1365-2265.2005.02339.x. PMID 16117815
- [Background] Isidori AM, Giannetta E, Gianfrilli D, Greco EA, Bonifacio V, Aversa A, Isidori A, Fabbri A, Lenzi A. Effects of testosterone on sexual function in men: results of a meta-analysis. Clin Endocrinol (Oxf). 2005 Oct;63(4):381-94. doi: 10.1111/j.1365-2265.2005.02350.x. PMID 16181230
- [Background] Isidori AM, Lenzi A. Testosterone replacement therapy: what we know is not yet enough. Mayo Clin Proc. 2007 Jan;82(1):11-3. doi: 10.4065/82.1.11. No abstract available. PMID 17285780
- [Background] Aversa A, Isidori AM, Spera G, Lenzi A, Fabbri A. Androgens improve cavernous vasodilation and response to sildenafil in patients with erectile dysfunction. Clin Endocrinol (Oxf). 2003 May;58(5):632-8. doi: 10.1046/j.1365-2265.2003.01764.x. PMID 12699447
- [Background] Aversa A, Isidori AM, De Martino MU, Caprio M, Fabbrini E, Rocchietti-March M, Frajese G, Fabbri A. Androgens and penile erection: evidence for a direct relationship between free testosterone and cavernous vasodilation in men with erectile dysfunction. Clin Endocrinol (Oxf). 2000 Oct;53(4):517-22. doi: 10.1046/j.1365-2265.2000.01118.x. PMID 11012578